CLINICAL TRIAL: NCT02399111
Title: A Prospective Randomized Control Trial to Evaluate Negative Pressure Incision Management System for Groin Wounds in Vascular Surgery Patients
Brief Title: A Trial to Evaluate Negative Pressure Incision Management System for Groin Wounds in Vascular Surgery Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI Decision
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Kambhampaty Krishnasastry, MD, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 13-485
Record Dates: First submitted 2015-02-24; First posted 2015-03-26 (Estimated); Results first posted 2016-11-21 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: Surgical Procedure, Unspecified
Keywords: Prevena Incision Management System (PIMS); Surgical Site Infection (SSI)
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Not obese:BMI<30; Standard Care (No Intervention): Standard Wound Care
- Obese:BMI≥30; Standard Care (No Intervention): Standard Wound Care
- Not Obese:BMI<30; Wound Vac (Other): Using Prevena Incision Management System
  Interventions: Device: Prevena Incision Management System
- Obese:BMI≥30; Wound Vac (Other): Using Prevena Incision Management System
  Interventions: Device: Prevena Incision Management System

INTERVENTIONS:
Device: Prevena Incision Management System — The PIMS unit is a single patient use, battery-powered, disposable unit that delivers continuous negative 125 mmHg pressure to the closed surgical incision for a 7-day therapy period. It is an easy to use device that also provides audible and visual alerts for low battery, maximum canister volume, and leak conditions. Additional alerts include system error and device life-cycle expiration (8 days). It is contained in a water-resistant housing, which allows the Subject to lightly shower with the device. Wound fluids are contained within the 45 mL canister. For the purposes of this clinical investigation, canisters can be replaced as often as is needed. A carrying case is also provided with the therapy unit, to allow for patient mobility during the therapy period.
  Arms: Not Obese:BMI<30; Wound Vac; Obese:BMI≥30; Wound Vac

SUMMARY:
The purpose of this research study is to investigate if a new negative pressure incision (surgical cut) management system, could reduce the occurrence of groin wound infections after vascular surgery. This is a single use, sterile dressing that is applied to the patient's skin. It has an attached battery-powered unit that provides negative pressure (a vacuum environment) to the dressing and a disposable canister for the collection of wound fluids. The patient is being asked to participate in this study because the patient is planning to have a vascular surgery procedure that involves groin incision.

DETAILED DESCRIPTION:
Surgical site infection (SSI) in groin wounds after vascular surgery is a significant contributing factor for increased morbidity. Despite the use of prophylactic systemic antibiotics, postoperative groin wound infection still occurs in some circumstances and it continues to be a serious problem after vascular surgical procedures. The incidence of SSI varies from 5 - 40%, and depending upon the depth of infection and type of vascular procedure, the morbidity could range from prolonged hospital stay to limb loss.

Increased incidence of SSIs in patients is related to systemic factors like Diabetes, hypertension (HTN), history of smoking, chronic obstructive pulmonary disease (COPD), and local factors like disruption of lymphatics, groin proximity to the perineum, previous surgery at the same site and the use of prosthetic graft material.

Prophylactic systemic antibiotics have been routinely used in all vascular surgery procedures, and despite of gentle tissue handling, proper hemostasis and other technical points to minimize tissue trauma, SSIs do happen.

The investigators hypothesize that using a closed dressing system with negative pressure will keep the surgical site protected from nearby contaminated field and decrease the risk of infection

ELIGIBILITY:
Inclusion Criteria:

1. Older than 18 years
2. Subjects are capable of giving informed written consent
3. Undergoing a vascular surgery procedure that involves a groin incision at North Shore University Hospital and Long Island Jewish Hospital.

Exclusion Criteria:

1. The patient has a history of blood clotting disorders
2. Patient has evidence of infection in the groin area, where surgical procedure is planned
3. Patient body habitus precludes placement of Prevena dressing.
4. Allergy to Silver or acrylic adhesive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kambhampaty Krishnasastry, MD, Principal Investigator — Northwell Health
Locations (1):
- North Shore-LIJ Health System, Lake Success, New York, United States

REFERENCES:
- [Background] Matatov T, Reddy KN, Doucet LD, Zhao CX, Zhang WW. Experience with a new negative pressure incision management system in prevention of groin wound infection in vascular surgery patients. J Vasc Surg. 2013 Mar;57(3):791-5. doi: 10.1016/j.jvs.2012.09.037. Epub 2013 Jan 9. PMID 23312938
- [Background] Colli A, Camara ML. First experience with a new negative pressure incision management system on surgical incisions after cardiac surgery in high risk patients. J Cardiothorac Surg. 2011 Dec 6;6:160. doi: 10.1186/1749-8090-6-160. PMID 22145641

RESULTS

PARTICIPANT FLOW:
Groups:
- Not Obese:BMI<30; Standard Care: Not obese: BMI< 30; Standard Wound Care
- Obese:BMI≥30; Standard Care: Obese: BMI ≥30; Standard Wound Care
Period: Overall Study
Arm/Group | Not Obese:BMI<30; Standard Care | Obese:BMI≥30; Standard Care | Not Obese:BMI<30; Wound Vac | Obese:BMI≥30; Wound Vac
Started | 4 | 1 | 4 | 0
Completed | 4 | 1 | 4 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Not Obese:BMI<30; Standard Care: Not obese:BMI<30;Standard Wound Care
- Obese:BMI≥30; Standard Care: Obese:BMI≥30;Standard Wound Care
- Total: Total of all reporting groups
Arm/Group | Not Obese:BMI<30; Standard Care | Obese:BMI≥30; Standard Care | Not Obese:BMI<30; Wound Vac | Obese:BMI≥30; Wound Vac | Total
Number analyzed (Participants) | 4 | 1 | 4 | 0 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 1 | 4 | 0 | 9
  >=65 years | 0 | 0 | 0 | 0 | 0
Gender [Count of Participants; unit: Participants]
  Female | 2 | 1 | 0 | 0 | 3
  Male | 2 | 0 | 4 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Wound Infection With Szilagyi Grade
Description: This study was terminated prior to gathering of data.
Time Frame: 30 days
Arm/Group | Not Obese:BMI<30; Standard Care | Obese:BMI≥30; Standard Care | Not Obese:BMI<30; Wound Vac | Obese:BMI≥30; Wound Vac
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: Assess the Safety of the Devise by Monitoring Incidence of Bleeding , Seroma Formation
Description: This study was terminated prior to collection of data.
Time Frame: 30 days
Arm/Group | Not Obese:BMI<30; Standard Care | Obese:BMI≥30; Standard Care | Not Obese:BMI<30; Wound Vac | Obese:BMI≥30; Wound Vac
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Not Obese:BMI<30; Standard Care | Obese:BMI≥30; Standard Care | Not Obese:BMI<30; Wound Vac | Obese:BMI≥30; Wound Vac
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/1 | 0/4 | 0/0
Other Adverse Events (participants affected / at risk) | 1/4 | 1/1 | 0/4 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Not Obese:BMI<30; Standard Care (N=4) | Obese:BMI≥30; Standard Care (N=1) | Not Obese:BMI<30; Wound Vac (N=4) | Obese:BMI≥30; Wound Vac (N=0)
Infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No